CLINICAL TRIAL: NCT01860339
Title: Growth and Development of Striatal-Cerebellum Circuitry in Subjects at Risk for Huntington's Disease
Brief Title: Child to Adult Neurodevelopment in Gene Expanded Huntington's Disease
Acronym: ChANGE HD
Status: Recruiting | Type: Observational
Sponsor: Peggy C Nopoulos (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Peggy C Nopoulos, Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 200507759; 2U01NS055903-10 (NIH)
Record Dates: First submitted 2013-05-16; First posted 2013-05-22 (Estimated); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Huntington's Disease
Keywords: Huntington's Disease; HD; Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Bio-specimens are collected and retained for all participants for genetic testing purposes and future research. Specimens are a single sample of 3-4 teaspoons of blood drawn from the arm. Optional saliva sample collection will be offered if unable to collect sufficient blood sample.
  Biospecimens will be tested for the number of CAG repeats in the Huntingtin Gene. Each sample obtained will be coded with a randomly assigned number and never linked with personal identifiers. The results from the genetic analysis will be sent directly to the data manager on the project, who is the ONLY research member with access to this data. This person has no direct contact with study participants.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Gene-expanded (GE): Children at risk for HD who have a CAG repeat length of 40 and above.
- Gene Non-Expanded (GNE): Children at risk for HD who have a CAG repeat length of 39 or less

SUMMARY:
Huntington's Disease (HD) is an autosomal dominant disease manifested in a triad of cognitive, psychiatric, and motor signs and symptoms. HD is caused by a triplet repeat (CAG)expansion in the gene Huntingtin (HTT). This disease has classically been conceptualized as a neurodegenerative disease. However, recent evidence suggests that abnormal brain development may play an important role in the etiology of HD. Huntingtin (HTT)is expressed during development and through life. In animal studies, the HTT gene has been shown to be vital for brain development. This suggests that a mutant form of HTT (gene-expanded or CAG repeats of 40 and above) would affect normal brain development. In addition, studies in adults who are gene-expanded for HD, but have not yet manifested the illness, (pre-HD subjects) have significant changes in the structure of their brain, even up to 20 years before onset of clinical diagnosis. How far back these changes are evident is unknown. One possibility is that these brain changes are present throughout life, due to changes in brain development,though initially associated with only subtle functional abnormalities.

In an effort to better understand the developmental aspects of this brain disease, the current study proposes to evaluate brain structure and function in children, adolescents, and young adults (ages 6-30) who are at risk for developing HD - those who have a parent or grandparent with HD. Brain structure will be evaluating using Magnetic Resonance Imaging (MRI) with quantitative measures of the entire brain, cerebral cortex, as well as white matter integrity via Diffusion Tensor Imaging. Brain function will be assessed by cognitive tests, behavioral assessment, and physical and neurologic evaluation. Subjects that are gene-expanded (GE) will be compared to subjects who are gene non-expanded (GNE). Changes in brain structure and/or function in the GE group compared to the GNE group would lend support to the notion that this disease has an important developmental component.

ELIGIBILITY:
Inclusion Criteria:

* Family history of Huntington's Disease
* Age 6-30 years
* Age-appropriate knowledge of HD and personal risk

Exclusion Criteria:

* Metal in body, including braces
* History of head trauma, brain tumor, seizures, epilepsy
* History of major surgery and/or significant ongoing medical issue(s)

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Young people ages 6-30 years old who have a parent or grandparent that has been diagnosed with Huntington's Disease
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2005-07 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Volume of brain structures as measured by Magnetic Resonance Imaging (MRI) | 1 hour out of 6-7 hour testing day, 3-4 annual visits
  Magnetic Resonance Imaging (MRI) and Diffusion Tensor Imaging (DTI) data will be analyzed to assess brain structure based upon variables including global volume, total cerebral spinal fluid, subregion volumes, cortical surface anatomy including cortical depth, surface area and gyral shape, and symmetry between brain hemispheres, all in consideration of age, gender, and height. Results will be evaluated for comparative differences between the GE group and the GNE group. In addition, these measures of brain structure will be paired with corresponding measures of brain function to evaluate brain development based upon growth and performance.

SECONDARY OUTCOMES:
Quantitative assessment of cognitive skills and behavioral factors | 4 hours out of 6-7 hour testing day, 3-4 annual visits
  Participants undergo a cognitive battery which will quantify skills such as attention, learning, memory. In addition, behavioral measures will be administered in both self and proxy report formats. Results will be analyzed for comparative differences between the GE group and the GNE group. In addition, these measures of brain function will be paired with appropriate measures of brain structure to evaluate brain development based upon growth and performance.

OTHER OUTCOMES:
Quantitative assessment of motor performance | 1 hour out of 6-7 hour testing day, 3-4 annual visits
  Motor skill (both fine and gross) will be assessed and quantified via standard UHDRS motor exam and Q-Motor/Q-Cog equipment suite. Results will be analyzed for comparative differences between the GE group and the GNE group. In addition, these measures of brain function will be paired with appropriate measures of brain structure to evaluate brain development based upon growth and performance.
Quantification of Neurofilament Light | 10 minutes for blood draw out of 6-7 hour testing day, 3-4 annual visits
  Plasma samples will be sent for each visit to University College of London for analysis of NfL, an indicator of neuronal damage, to determine viability as a biomarker for Huntington's Disease.

CONTACTS AND LOCATIONS:
Overall Officials: Peggy C Nopoulos, MD, Principal Investigator — University of Iowa
Locations (6):
- United States (6):
  - University of California Davis, Sacramento, California
  - University of Iowa Hospitals and Clinics, Department of Psychiatry, Iowa City, Iowa
  - Columbia University Medical Center, New York, New York
  - Children's Hospital of Philadelphia with the University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Aggregate, de-identified data may be shared with approved collaborators, but individual participant data will not be shared.

REFERENCES:
- See also: Previous study site — http://www.kids-hd.org
- See also: Facebook page — https://www.facebook.com/ChangeHDresearch/
- See also: Twitter account — https://twitter.com/ChANGEHD_study